CLINICAL TRIAL: NCT06728319
Title: A Multicenter, Retrospective, Chart Review Study Evaluating the Impact and Utility of the Blood-Based Proteomic Integrated Classifier and Auto-Antibody Tests in the Real-World
Acronym: CLARIFY
Status: Active, not recruiting | Type: Observational
Sponsor: Biodesix, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BDSX-CD-011
Record Dates: First submitted 2024-10-04; First posted 2024-12-11 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Lung Nodules
Keywords: Lung nodule; Pulmonology

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a multicenter retrospective chart review. Sites with at least 100 patients tested with the IC and AAT tests, who have index dates (date of IC and AAT testing) at least one year prior to data collection date will be eligible for participation.

DETAILED DESCRIPTION:
This study is a multicenter retrospective chart review. Sites with at least 100 patients tested with the IC and AAT tests, who have index dates (date of IC and AAT testing) at least one year prior to data collection date will be eligible for participation.

The protocol will require institutional IRB approval and a waiver of patient consent will be obtained. The data to be collected will be de-identified when entered into the study database. The collection of this de-identified data does not pose any risk to the subjects and does not require any further testing of the patient. The chart review will utilize a third-party Clinical Research Associate (CRA) with certified ICH-GCP training for data collection and documentation. Biodesix, Inc. in conjunction with the CRA will develop and maintain the Electronic Data Capture (EDC) system.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated at sites with ≥100 patients who have been evaluated with the IC and AAT tests.
* Patients who are at least 40 years of age on the index date.
* Patients who have index dates (date of IC and AAT testing) at least one year prior to data collection date.

Exclusion Criteria:

* Patients with no prior AAT and/or IC testing at the study site.
* Patients less than 40 years of age on the index date.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that have previously been tested with the AAT and IC tests and have at least 1 year of follow up data.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Assess Test Performance of AAT test | Up to 24 months
  To assess the performance of the AAT test in a real-world patient population:
  1. Sensitivity of the AAT test at 24 months
  2. Specificity of the AAT test at 24 months
  3. Positivity predictive value of the AAT test at 24 months
Assess Test Performance of IC test | 24 months
  To assess the performance of the IC test in a real-world population:
  1. Sensitivity of the IC test at 24 months
  2. Specificity of the IC test at 24 months
  3. Negative predictive value of the IC test at 24 months
Assess serial performance of serial testing with the AAC and IC tests. | 24 months
  Assess the performance of the of serial testing with the AAC and IC tests

SECONDARY OUTCOMES:
Assess ATT Test Accuracy | Up to 24 months
  To assess the accuracy of the AAT post-test risk of malignancy by comparing with the actual patient outcome.
  * Compare the AAT test predicted proportion of malignant nodules to the actual proportion of malignant nodules by probability decile.
  * Compare the IC test predicted proportion of malignant nodules to the actual proportion of malignant nodules by probability decile.
Determine Health Outcomes | Up to 24 months
  To determine one-year health outcomes of patients stratified by AAT and IC tests result risk categories.
  * The number and type of invasive diagnostic procedure performed on newly identified nodules stratified by AAT test results.
  * The number of patients routed to CT surveillance following initial nodule evaluation that result in nodule resolution or up to 24-month radiographic stability stratified by the AAT test.
  * The number and type of invasive diagnostic procedures performed on newly identified nodules stratified by IC test results.
  * The number of patients routed to CT surveillance following initial nodule evaluation that result in nodule resolution or up to 24-month radiographic stability stratified by the IC test.
  * The number of malignant nodules identified following a diagnostic procedure stratified by histology and stage.
  * The number of specific benign nodules identified following a diagnostic procedure, stratified by pathological findings.

OTHER OUTCOMES:
Assess Test Performance in Sub-Populations | Up to 24 months
  Assess the performance of the AAT and IC tests in patient subpopulations.
  1. Sensitivity of the AAT test in patient sub-populations at 24 months
  2. Specificity of the AAT test in patient sub-populations at 24 months
  3. Positivity predictive value of the AAT in patient sub-populations test at 24 months
  4. Sensitivity of the IC test in patient sub-populations at 24 months
  5. Specificity of the IC test in patient sub-populations at 24 months
  6. Negative predictive value of the IC test in patient sub-populations at 24 months
Assess Test Performance in Populations Outside of Validation | Up to 24 months
  To assess the performance of the AAT and IC tests in populations outside of their primary validated populations.
  1. Sensitivity of the AAT test in patient sub-populations at 24 months
  2. Specificity of the AAT test in patient sub-populations at 24 months
  3. Positivity predictive value of the AAT in patient sub-populations test at 24 months
  4. Sensitivity of the IC test in patient sub-populations at 24 months
  5. Specificity of the IC test in patient sub-populations at 24 months
  6. Negative predictive value of the IC test in patient sub-populations at 24 months

CONTACTS AND LOCATIONS:
Overall Officials: James Jett, MD, Principal Investigator — Biodesix, Inc.
Locations (5):
- United States (5):
  - Pulmonary & Sleep of Tampa Bay, Brandon, Florida
  - White-Wilson Medical Center, Fort Walton Beach, Florida
  - The Lung and Sleep Disorder Institute, Somerset, Kentucky
  - Southcoast Health System, Fairhaven, Massachusetts
  - The Lung Center, PC, DuBois, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor website — https://www.biodesix.com/